CLINICAL TRIAL: NCT04796870
Title: Outcomes of Powerbraining: the RHBS Brain and Balance Study of Older Adults
Brief Title: RHBS Brain and Balance Study of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Powerbraining
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Cognitive Performance; Balance
Keywords: Attention; Working Memory; Visual Spatial Memory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Online Brain and Balance Training (Experimental): Individuals that meet the inclusion/exclusion criteria and enrolled in the study will participate in a 8-week virtual balance and cognitive training intervention performed three times a week.
  Interventions: Other: Online Brain and Balance Training Program

INTERVENTIONS:
Other: Online Brain and Balance Training Program — The intent of the intervention is to encompass cardiovascular conditioning, cognitive performance and balance performance improvements. To promote cardiovascular conditioning the exercises are structured to keep the participant in motion while maintaining an elevated heart rate using techniques such as squats, marching and upper extremity movements. The video provides adaptations to increase or decrease the challenge based on subject ability. To promote cognitive performance, participants will be asked to complete simple and complex cognitive tasks, such as arithmetic, spatial memory recall and attention while completing the physical exercises. To promote balance performance, the videos include single limb stance and weight shifting tasks. Videos are presented in a progressively challenging manner for all domains.

SUMMARY:
Brief Summary:

Cognition and balance are known to decline during the aging process. Cognitive performance is essential for functional independence and determines whether an individual can perform instrumental daily living activities (e.g., finances, driving, independent living). Balance is critical for participation in everyday life activities. Impaired balance increases fall risk, and subsequent injury increased caregiver dependency and decreased independence.

The purpose of this study is to investigate the outcomes of 24 sessions of online mobility and cognitive training (35 minutes/session, 3x/week, 8-12 weeks) for community-based older adults. The exercise program is progressively challenging and emphasizes balance, cardiovascular conditioning, attention, and working memory. The primary outcomes of interest are cognitive performance and balance changes, with secondary outcomes relating to self-efficacy, resilience, and physical activity.

DETAILED DESCRIPTION:
Protocol Overview: Subjects will be recruited from the greater Washington D.C. metro area. Individuals interested in participating as subjects will complete initial verbal screening to determine eligibility for inclusion. Those subjects who volunteer to participate will then be consented and enrolled for participation if exclusion and inclusion criteria are met.

Visit 1: (~120 minutes) Participants meeting study rationale and voluntarily agree to participate will receive a standardized email generated through the Research Electronic Data Capture (REDcap) platform. The email will contain a Zoon videoconference link to complete cognitive assessments (described below) and virtual balance tests (described below) with a research assistant. That email will also contain a second link to complete all surveys through the REDcap portal. Only one selected member of the research team will have an identification key connecting personally identifiable information to returned surveys. Cognitive assessments will be completed online using REDcap and Q-global Pearson, with a member of the research team providing verbal instruction via videoconference. After cognitive assessment completion, participants will perform the virtual balance tests. A team member will oversee setup via videoconference to ensure the environment's safety and administer the test. Participants will receive login instructions and access code to the virtual training sessions with POWER BRAINing.

Visits 2-25: (~35 minutes each) Participants will perform training videos at their convenience two to three times per week for 8-12 weeks for a total of 24 sessions. Participants will receive a weekly email and/or phone call from research staff to check safety, provide encouragement, and answer any questions.

Visit 26: (~120 minutes) Subjects will repeat the same testing procedures, in the same order, as they did in visit 1.

Study Procedures:

Cognitive Outcome Measures: The following assessments will be administered via videoconference using the Zoom platform, and data will be stored in REDcap. Directions will be given verbally using the specified script for each outcome measure.

Digit Span subset of Wechsler Adult Intelligence Scale- 4th Edition (WAIS-IV, 10 minutes): Digit Span, which has two subsections forward (DS-F) and backward (DS-B), evaluates attention and auditory working memory respectfully. The DS-F requires participants to repeat numbers in the same order as they were read aloud by the examiner. The testing administrator will say to the subject, "I am going to read you a sequence of digits, and I want you to try and repeat the digits in the same order they were read out loud." To minimize confusion, this example will be provided, "If I say '4, 7, 1', then you would repeat those same digits in that same order". The DS-B requires participants to repeat the numbers in reverse order of what was presented aloud by the examiner. The test administrator will say, "I am going to read you a sequence of digits, and I want you to try and repeat the digits in the reverse order they were read out loud. For example, if I say '4, 7, 1', then you would repeat those same digits backward." In both subsets, the sequences increase in length as the participant progresses, each length has two different sequences. The DS-F has 16 sequences, and the DS-B has 14 sequences. The maximum raw score of DS-F is 16 and DS-B is 14. The digits will be read in an even tone, at approximately the rate of one digit per second. The first set of sequences will begin at three digits. The discontinuation criterion is the failure to reproduce two sequences of equal length correctly.

Letter-Number Sequencing (LNS, 5 minutes): The LNS requires participants to listen to a series of number and letter and repeat the sequence starting first with the numbers in ascending order, followed by the letters in alphabetical order. The testing administrator will say to the subject " "I am going to say a set of numbers and letter. Your task is report them by first saying the numbers in ascending order and then the letters in alphabetical order. For example, if I say '9, T, 3, A', your response would be '3, 9, A, T'." The numbers and letters will be read in an even tone, at approximately the rate of one digit/number per second. The first sequence begins at two and increases in length as the participant progresses. The maximum raw score is 21. Discontinuation criterion is failure to correctly reproduce three sequences of equal length.

Simple and Choice Reaction Time (10 minutes): The simple (SRT) and choice (CRT) response time tasks record reaction time to measure the speed of information processing using an online visual stimulus task. The participant will begin with the SRT and will be asked to "Wait until you see a black 'X' in the white square. When that happens, press the spacebar. The goal is to respond as quickly as possible". In the CRT task, there are four possible stimuli and four possible stimulus-response associations. Directions are as follows, "Wait until you see a black 'X' in one of the four white squares. When that happens, press the corresponding key (z, x, <or >). You can use both hands and may keep your fingers on the keys throughout the test. The goal is to respond as quickly as possible". The participant will have one practice round for each task.

Spatial Addition subset of Wechsler Memory Scale- 4th Edition (WMS-IV, 15 minutes): This subtest examines visual-spatial working memory and will be administered using the Q-global Pearson platform. The participant is shown two 4x4 grids for five seconds each. Both stimuli will contain blue dots, red dots, or both. The participant must memorize the dots' color and location in each stimulus to create a final grid that adds the blue dots' locations, ignores any red dots, and subtracts the location of blue dots that overlap. The instructions will include: "In this next task, you will be shown two grids for 5 seconds each that contain red or blue dots. Your task in the third grid is to create a final grid that adds the spatial location of the blue dots, subtracting any blue dots that overlapped and ignore any red dots". Participants will be shown an example of this task.

Balance outcome measures: The following assessments will be performed via videoconference using Zoom with a research team member who will oversee the participants' setup for optimal safety and visualization. The participant will be cued to prioritize safety, upright balance during tests. Participants are encouraged to position themselves with the back of a chair, a countertop, or a wall within reach to their front or side, as they perform these tests. The virtual test administrator will ensure a safe environment before starting the test.

30-second Chair Stand (~5 minutes): A test of leg strength where the number of times a participant can stand up fully and sit back down within 30 seconds with arms crossed over their chest. Ideally, the chair has a straight back that does not have armrests and, ideally, without armrests with the seat seventeen inches above the floor. Most importantly for this assessment is using the same chair during pre- and post-assessments. Participants will place the chair against a wall to ensure it will not move. Ideally, camera orientation is lateral to the participant to verify achieving full stand and sit for each repetition and not bracing knees/legs against the chair. Participants must use the same chair during baseline and follow-up testing.

Four-Stage Balance Test (~10 minutes): The purpose is to assess static balance in a standing position without using an assistive device. Patients will balance with their feet in four positions that get progressively more challenging. Positions include feet together, staggered, heel-to-toe, and single leg. Participants will stand up to 10 seconds in the first three positions and up to 30 seconds while in a single leg stance to minimize a ceiling effect. The participant may adjust their arms to maintain balance, but the test is over if they grab a support surface or changes foot-position. Test administrator times each position stance when the participant achieves the testing position without UE support. If the person holds a position for 10 seconds without moving their feet or needing support, that position is complete, and the participant returns to a bilateral stance. If the participant cannot hold the position for 10 seconds, the time is over, and the sustained time is documented (i.e., the participant does not progress to the next test position). The final position (single-limb stance) is held for up to 30 seconds, with documentation of the length of time held in seconds.

Questionnaires:

Screening Tool: This questionnaire is study-specific, developed to assess the eligibility criteria of inquiring individuals and provide standardized information on the purpose of this study. It is administered by research staff via phone call and recorded in the REDcap platform.

Testing/Forms:

Physical Activity Readiness Questionnaire (PAR-Q, 5 minutes): The PAR-Q is a 7 question screening tool used to assess an individual's physical fitness level and ability to engage in physical activity. The PAR-Q will be administered in REDcap after meeting the criteria via phone screening.

Connor Davidson Resilience Scale (~10 minutes): The Connor Davidson Resilience Scale is a one-dimensional self-reported scale consisting of 25 items measuring resilience and will be administered through an online survey REDcap on visit-1 and visit 26.

Activities-Specific Balance Confidence Scale (ABC Scale, 5-10 minutes): The ABC scale is a 16-item self-report rating confidence in performing various activities. The ABC Scale will be administered through an online survey through REDcap on visit-1 and visit-26.

Outpatient Physical Therapy Improvement in Movement Assessment Log (OPTIMAL, 20 minutes): The OPTIMAL scale measures self-confidence and difficulty performing 21 functional activities and will be administered through an online survey through REDcap on visit-1 and visit-26.

International Physical Activity Questionnaire- Long Form (~15-30 minutes): The IPAQ is a 27-item self-reported measure of physical activity to compare levels between populations internationally. It will be administered through an online survey through REDcap on visit-1 and visit-26.

Online Video Intervention: The intervention intends to encompass cardiovascular conditioning, cognitive performance, and balance performance improvements. The exercises are structured to keep the participant in motion to promote cardiovascular conditioning while maintaining an elevated heart rate using techniques such as squats, marching, and upper extremity movements. The video provides adaptations to increase or decrease the challenge based on subject ability. Participants will be asked to complete simple and complex cognitive tasks to promote cognitive performance, such as arithmetic, spatial memory recall, and attention while completing the physical exercises. The videos include single-limb stance and weight shifting tasks to promote balance performance. Videos are presented in a progressively challenging manner for all domains.

ELIGIBILITY:
Inclusion Criteria:

* 55 - 80 years old
* Ability to take at least 4 steps without an assistive device
* Ability to speak English

Exclusion Criteria:

* Inability to ambulate at least 4 steps without assistive device
* Uncontrolled cardiovascular, pulmonary, neurological, or metabolic disease which may impact the ability to exercise or in which exercise is contraindicated
* Cognitive or psychiatric impairment precluding informed consent or ability to following instructions

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Change in Attention and Auditory Working Memory | pre and post 8-week intervention protocol
  (A) as measured by the Digit Span subset of Wechsler Adult Intelligence Scale- 4th Edition (WAIS-IV); Each correct response is worth 1 point, with a maximum of 14 for each sub-score and for a total score of 24. Higher scores are indicative of better outcome. (B) as measured by Letter-Number Sequencing, each correct response is worth 1 point, with a maximum total score of 21. Higher scores are indicative of better outcome.
Change in Visual Spatial Working Memory | pre and post 8-week intervention protocol
  as measured by the Spatial Addition Subset of Wechsler Memory Scale- 4th Edition (WMS-IV); This is a 24-item assessment, each correct response is worth 1 point for a total score of 24. Higher scores are indicative of better outcome.
Change in Information Processing Speed | pre and post 8-week intervention protocol
  as measured by the Simple and Choice Reaction Times
Change in Static Balance in a Standing Position | pre and post 8-week intervention protocol
  as measured by the Four-Stage Balance Test

SECONDARY OUTCOMES:
Change in Resilience | pre and post 8-week intervention protocol
  as measured by the Connor Davidson Resilience Scale. This is a 25 item assessment. Scoring of the scale is based on summing the total of all items, each of which is scored from 0-4.The full range is from 0 to 100, with higher scores reflecting greater resilience.
Change in Confidence in Performing Various Activities | pre and post 8-week intervention protocol
  as measured by the Activities-Specific Balance Confidence Scale; The ABC is an 11-point scale and ratings should consist of whole numbers (0-100) for each item. Total the ratings (possible range = 0 - 1600) and divide by 16 to get each subject's ABC score. Higher score is indicative of better confidence.
Change in Level of Physical Activity | pre and post 8-week intervention protocol
  as measured by the International Physical Activity Questionnaire- Long Form; Results can be reported in categories (low activity levels, moderate activity levels or high activity levels). Scoring a HIGH level means your physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level. Scoring a MODERATE level means you are doing some activity more than likely equivalent to half an hour of at least moderate intensity physical activity on most days. Scoring a LOW level means that you are not meeting any of the criteria for either MODERATE of HIGH levels of physical activity.
Change in Leg Strength | pre and post 8-week intervention protocol
  as measured by the 30-second Chair Stand Test
Change in Lower Extremity Kinematic parameters | pre and post 8-week intervention protocol
  as measured during the 30-second Chair Stand
Change in Postural Sway | pre and post 8-week intervention protocol
  as measured during the Four-Stage Balance Test

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Guccione, PT, PhD, DPT, Principal Investigator — George Mason University
Locations (1):
- George Mason University, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No